CLINICAL TRIAL: NCT07186556
Title: Cancer-related Fatigue and Its Biological Contributors in Adolescent and Young Adult Brain Tumor Survivors: Effects of a Tele-exercise Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-1036; NCI-2025-06748 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Fatigue; Brain Tumor Adult
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control Group (Experimental): Participants will randomized using incorrect baseline information.
  Interventions: Behavioral: RISE-YA Intervention
- InItervention Group: Remote Implementation of Supervised Exercise for Young Adult (Experimental): Participants will randomized using incorrect baseline information.
  Interventions: Behavioral: Survivorship Education

INTERVENTIONS:
Behavioral: RISE-YA Intervention — Participants will receive energy conservation (EC) counseling, behavior coaching, and exercise training.
  Arms: Attention Control Group
Behavioral: Survivorship Education — During weeks 1-6 and 1 time a week during Weeks 7-12, participants will receive a video call which will last about 60 minutes.
  Arms: InItervention Group: Remote Implementation of Supervised Exercise for Young Adult

SUMMARY:
The goal of this research study is to learn about the effects of the RISE-YA intervention on cancer-related fatigue in young adults who are brain cancer survivors.

DETAILED DESCRIPTION:
Primary Objective:

Test the efficacy of RISE-YA to improve CRF

Secondary Objectives:

1. Test the efficacy of RISE-YA to improve PA and physical function in fatigued YA brain tumor survivors.
2. Determine A) cross-sectional associations of CRF with oxidative phosphorylation (OxPhos) and with inflammation, and B) the effect of RISE-YA on OxPhos and on inflammation.

Exploratory Objective:

Assess the effect of our supervised exercise intervention on patient-reported health-related quality of life, muscle mass development (BMI, skinfold and circumferences [waist, arm, and calf area]), patient-reported dietary intake, and exercise adherence and progression.

ELIGIBILITY:
Inclusion Criteria:

1. Is currently between the ages of 18-39 years
2. Their primary brain tumor was diagnosed at age 15-39 years
3. Is 6 months to <5 years post curative treatment
4. Has been treated with chemotherapy and radiation, given most patients receive both therapies.
5. Functional Assessment of Chronic Illness therapy (FACIT)-Fatigue ≤ 43. FACIT-Fatigue will be used as a screener because this 13-item scale can be completed relatively quickly in clinic
6. Currently engage in <150 minutes of PA and < 2 sessions of muscle strengthening exercise per week (assessed by Godin Leisure-Time PA Questionnaire)
7. Must be able to speak, write, and read English
8. No exercise contraindication as assessed by screening with the Physical Activity Readiness Questionnaire PAR-Q+. In addition, participants' care teams will be notified of their participation in the study.
9. Must be able to provide informed consent/assent.

Exclusion Criteria:

1. Non-English speaking
2. Screen failure for exercise safety
3. Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease
4. Recent fracture or acute musculoskeletal injury that precludes ability to participate in supervised exercise training sessions
5. History of underlying chronic disease, secondary malignances, germline genetic syndrome, or recurrent disease requiring re-irradiation of the brain
6. Cognitive and/or major sensory deficits that would impede the completion of research activities and assessments as deemed by the clinical team.
7. Self-report of pregnancy
8. Prisoners
9. Documented developmental disorders (e.g., Autism) or major psychotic illness (e.g., schizophrenia)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roth, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org